CLINICAL TRIAL: NCT06408337
Title: Phase I-IIa, Randomized, Controlled, Open-label, Single-center Clinical Trial to Evaluate Safety, Feasibility, and Efficacy of the Use of BIOCLEFT in the Treatment of Patients With Cleft Palate
Brief Title: Phase I-IIa, to Evaluate the Safety, Feasibility, and Efficacy of the Use of BIOCLEFT in the Treatment of Cleft Palate.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Elisa María Cubiles Montero de Espinosa (Other)
Collaborators: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Responsible Party: Sponsor-Investigator, Elisa María Cubiles Montero de Espinosa, responsible for clinical trials, Fundación Pública Andaluza para la Investigación Biomédica Andalucía Oriental
Organization: Fundación Pública Andaluza para la Investigación Biomédica Andalucía Oriental (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIB-BIO-2023-03
Record Dates: First submitted 2024-04-25; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Cleft Lip and Palate
MeSH Terms: conditions — Cleft Lip | interventions — Drug Implants

STUDY DESIGN:
Intervention Model Description: The initial phase of the trial is non-randomized and involves the sequential recruitment of 5 subjects. All of them will be implanted with the autologous substitute for the human palatal mucosa of nanostructured fibrin-agarose generated by tissue engineering (BIOCLEFT), after reconstruction of the palate. In the second phase, the remaining patients (10) will be recruited, who will be randomized 1:1, so that 5 of these patients will be implanted with the investigational medication while undergoing standard surgical reconstruction. (uranostaphyllorrhaphy), while the other 5 will only undergo standard surgical reconstruction and will constitute the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): The experimental group will be implanted with an autologous human palatal mucosa substitute made of nanostructured fibrin-agarose generated by tissue engineering (BIOCLEFT). The implantation of this advanced therapy medication will cover the lateral defect generated by the mobilization of fibromucous flaps during standard surgery (uranostaphylorrhaphy
  Interventions: Procedure: implantation with an autologous human palatal mucosa substitute made of nanostructured fibrin-agarose generated by tissue engineering (BIOCLEFT).
- control group (No Intervention): These patients will be included in the control group and will receive the usual treatment for their disease (uranoestafilorrafia), without applying any type of restriction to the area used for the movement of the arms.

INTERVENTIONS:
Procedure: implantation with an autologous human palatal mucosa substitute made of nanostructured fibrin-agarose generated by tissue engineering (BIOCLEFT). — cleft palate repair surgery, all patients in the study will receive the standard treatment (uranostaphyllorrhaphy), with the only difference that patients assigned to the experimental study group will additionally have BIOCLEFT tissue obtained through tissue engineering grafted onto them. the lateral area of the palatine bone exposed when mobilizing the flaps. For the implant, the BIOCLEFT fabric will be placed in the area of exposed bone, sized to the size of the defect and sutured using uncoated, monofilament long-term absorbable synthetic suture.
  Arms: experimental

SUMMARY:
Phase I/II, controlled, open-label, randomized, single site clinical trial to assess the safety and feasibility, as well as hint efficacy evidence of a bioengineered palate mucosa substitute on nanostructured fibrin-agarose scaffolds with autologous mucosa tissue-specific cells (culture-expanded fibroblasts and keratinocytes), for tissue replacement and repair of donor area after the reconstruction of palate cleft defects (staphylorraphy), in comparison with standard care for donor mucosa.

DETAILED DESCRIPTION:
The initial phase of the trial is non-randomized, and involves the sequential recruitment of 5 eligible subjects with a minimum safety period of 30 days between them. All of them will be implanted with the autologous human palatal mucosa substitute of nanostructured fibrin-agarose generated by tissue engineering (BIOCLEFT), after reconstruction of the palate. Once the 5th treated patient has reached 1.5 months of follow-up after the intervention (Visit 8), the safety and feasibility data analysis will be carried out by the Independent Data Safety and Monitoring Committee (interim analysis), after which will allow continuation to the randomized phase of the trial, if the results allow it.

In the second phase, the rest of the patients (10) will be recruited, who will be randomized 1:1, such that 5 of these patients will be implanted with the investigational medication while undergoing standard surgical reconstruction. (uranostaphyllorrhaphy), while the other 5 will only undergo standard surgical reconstruction and will constitute the control group.

The total number of patients to be included in the study will be 15, who will be followed for 24 months according to a protocolized scheme that includes 2 pre-implant visits, 1 implant visit and 9 post-implant evaluation visits.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients, of both sexes.
* Diagnosis of total unilateral non-syndromic cleft lip and palate (FLPNS) that will undergo surgery for correction.
* Children who have previously donated a sample of oral mucosa during the cleft lip repair procedure (cheiloplasty).
* Informed consent signed by one or both parents (or legal guardian) adequately informed of the study and willing to follow the trial procedures and instructions.

Exclusion Criteria:

* Active infectious diseases.
* Allergies or hypersensitivity to any of the components/excipients of the Investigational Product.
* Severe hematological disorders/blood dyscrasias.
* Severe hepatic or renal dysfunction/failure.
* Serious endocrine disorders/dysfunctions.
* Malignant neoplasms
* Active HIV, HBV or HCV infection.
* Metabolic bone diseases (Paget's disease, hypercalcemia, etc.).
* Children with cleft lip and palate who present other congenital malformations that, in the opinion of the researcher, could affect the result of the study or the interpretation of the results of the study.
* Any other pathology that in the opinion of the investigator should not be included in the study for other medical or social reasons.

Ages: 10 Months to 14 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2028-04-17 (Estimated); Study Completion 2028-12-17 (Estimated)

PRIMARY OUTCOMES:
Evaluate implant´s feasibility and appearance of adverse events and serious adverse events related to treatment | 24 months
  Incidence of Serious Adverse Events after at the time of the implant of study drug.

SECONDARY OUTCOMES:
Evaluation of the time of the regeneration and healing of the lateral defect of the palatine bone from the moment of the intervention | 24 months
Evaluation of the aesthetic result through analysis of photographs | 24 months
  A scale designed ad hoc for the present trial will be used (aesthetic appearance assessment scale)
Preliminary evaluation of craniofacial growth through analysis of craniofacial photographs | 24 months
Hearing evaluation | 24 months
  Otoscopic/otomicroscopic examination and tympanogram by the otorhinolaryngologist, and placement of aeration tubes if considered necessary. The need or not to perform follow-up during the trial visits will be assessed depending on whether or not the patient presents any type of pathology.
Quality of life evaluation | 24 months
  Changes in quality of life will be assessed through the TAPQOL questionnaire for children between 1-5 years old.
Functional evaluation by the speech therapist | 24 months
  Evaluation of nasal escape; palate mobility; swallowing and articulation of functional language by the speech therapist.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Virgen de las Nieves, Granada, Spain/Granada, Spain

REFERENCES:
- [Derived] Espana-Lopez A, Fernandez-Valades R, Cubiles E, Garzon I, Martin-Piedra MA, Carriel V, Campos F, Martinez-Plaza A, Vallejo D, Liceras-Liceras E, Chato-Astrain J, Garcia-Garcia OD, Sanchez-Porras D, Avila-Fernandez P, Etayo-Escanilla M, Quijano B, Aguilar E, Campos A, Carmona G, Alaminos M. Phase I-IIa clinical trial to evaluate the safety, feasibility and efficacy of the use of a palate mucosa generated by tissue engineering for the treatment of children with cleft palate: the BIOCLEFT study protocol. BMJ Open. 2024 Dec 5;14(12):e093491. doi: 10.1136/bmjopen-2024-093491. PMID 39638596